CLINICAL TRIAL: NCT02920892
Title: Effects of AFQ056 on Language Learning in Young Children With Fragile X Syndrome (FXS)
Brief Title: AFQ056 for Language Learning in Children With FXS
Acronym: FX-LEARN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elizabeth Berry-Kravis (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Elizabeth Berry-Kravis, Professor of Pediatrics, Neurological Sciences, Biochemistry, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORA 15060903; 1U01NS096767-01 (NIH)
Record Dates: First submitted 2016-09-28; First posted 2016-09-30 (Estimated); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — mavoglurant

STUDY DESIGN:
Intervention Model Description: The trial will use a double-blind placebo-controlled parallel-group flexible-dose forced titration design. 100 eligible subjects with Fragile X Syndrome age 32 months to 6 years will enter a 4-month single-blind placebo lead-in period, followed by an 8-month double-blind treatment period during which subjects will randomized 1:1 to AFQ056 or placebo and will receive 6 months of language intervention. Subjects will then be invited to participate in an open-label extension phase during which all participants will receive treatment with active drug and continue language intervention for up to 8 months.
Who Masked: Participant, Investigator
Masking Description: After screening assessments, participants who met entry criteria and agreed to participate entered a single-blind 4-month placebo lead-in during which study participants had therapy treatments as usual to control for the effects of the language intervention. The 4-month placebo lead-in allowed for placebo effects to stabilize.
  At the end of the 4-month placebo lead-in, all participants will enter a double blind placebo controlled phase in which they will have a repeat battery of AFQ056 baseline assessments and will be randomized 1:1 to AFQ056 or placebo. Both treatment groups received an intensive language intervention for 6 months after 2 months of flexible dose titration to establish their maximum tolerated dose (MTD).
  After 8 months of treatment in the placebo-controlled phase (including 6 months of language intervention), all participants had final assessments and entered the open label extension (OLE) of about 8 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-Blind AFQ056 with language intervention (Experimental): After a 4-month single-blind placebo lead-in period, subjects with FXS were randomized to receive AFQ056 suspension by mouth twice per day in an 8 month double-blind treatment period.
  During the double-blind treatment period, subjects in the AFQ056 treatment group began with a dose of 25 mg AFQ056 twice per day and titrated to their maximum tolerated dose over the course of 7 weeks. After 7 weeks the dose was fixed, and at the 2 month visit, the intensive language intervention was initiated. Subjects continued the language intervention while remaining on a stable dose of AFQ056 (ranging from 12.5 mg BID to 100 mg BID), for the next 6 months.
  Safety and efficacy assessments were performed throughout.
  Interventions: Drug: AFQ056; Other: Language Intervention
- Double-Blind Placebo with language intervention (Placebo Comparator): After a 4-month single-blind placebo lead-in period, subjects with FXS were randomized to receive a placebo suspension by mouth twice per day in an 8 month double-blind treatment period.
  During the double-blind treatment period, dose titration to maximum tolerated dose of matching placebo occurred over 7 weeks. After 7 weeks, the dose was fixed, and at the 2 month visit, the intensive language intervention was initiated. Subjects continued the language intervention while remaining on placebo for the next 6 months.
  Safety and efficacy assessments were performed throughout.
  Interventions: Drug: Placebo; Other: Language Intervention
- Open-Label AFQ056 with language intervention (Experimental): After 8 months of treatment in the placebo-controlled phase, all subjects had assessments completed and were given the opportunity to enter the open-label extension (OLE) in which all subjects received AFQ056. The OLE began with 2 months of flexible dose titration to each subject's maximum tolerated dose followed by a period of stable treatment. Subjects also continued the language intervention through the extension phase.
  The duration of the stable treatment depended on when the subject was enrolled into the study. Those enrolled prior to June 15-30, 2019 received a 6-month period of stable treatment. Those enrolled after June 15, 2019 had their period of stable treatment shortened on a sliding scale, such that their treatment including weaning, if necessary, ended before August 31, 2021 (study drug expiration).
  Interventions: Drug: AFQ056; Other: Language Intervention

INTERVENTIONS:
Drug: AFQ056 — 12.5 mg - 100 mg oral suspension (liquid)
  Other Names: Mavoglurant
  Arms: Double-Blind AFQ056 with language intervention; Open-Label AFQ056 with language intervention
Drug: Placebo — Placebo oral suspension (liquid)
  Arms: Double-Blind Placebo with language intervention
Other: Language Intervention — All subjects will begin an intensive language intervention 2 months after starting treatment with AFQ056 or placebo and will continue the intervention through the end of the study.
  The language intervention will be administered by a trained language specialist through a combination of in clinic visits and at home synchronous video conferencing sessions. The intervention will subsequently be delivered to the parent by a speech-language clinician through weekly clinician coaching, homework, and feedback sessions.
  The language intervention is designed to help parents learn and use verbally responsive interactional strategies more frequently and effectively throughout the course of their daily interactions with their children.

SUMMARY:
The purpose of this clinical trial is to investigate the impact of AFQ056 on language learning in 3-6 year old children with Fragile X Syndrome (FXS).

DETAILED DESCRIPTION:
This study will enroll 100 participants with Fragile X syndrome (FXS) between the ages of 32 months and 6 years.

After being informed about the study and its potential risks, patients with Fragile X Syndrome will be screened for eligibility. Participants who meet entry criteria and agree to participate will then enter a single-blind 4-month placebo lead-in during which study participants will continue therapy treatments as usual to allow for placebo effects to stabilize. At the end of the 4-month placebo lead-in, all participants will have a repeat battery of AFQ056 baseline assessments and will enter the placebo-controlled phase, where they will be randomized in a 1:1 ratio to AFQ056 or placebo. All subjects will begin at a dose of 25 mg of AFQ056 or placebo, taken orally twice per day. Over 7 weeks, they will titrate up to their maximum tolerated dose (MTD), up to 100 mg. Once they have reached their MTD, both participant groups will initiate an intensive language intervention designed to maximize the extent to which parents engage in types of verbally responsive interactions that have been well documented as facilitating language learning. The entire language intervention will be delivered to the parent in the home or at scheduled study visits through the use of a laptop computer equipped with distance video-teleconferencing software and will include coaching, homework, and feedback sessions. Subjects will be treated with their MTD in combination with the language intervention for 6 months.

After 8 months of treatment in the placebo-controlled phase (including 6 months of language intervention), all participants will have final assessments and will be given the opportunity to enter the open label extension (OLE) period. In the OLE, all participants will be treated with active drug according to the same schedule as in the placebo-controlled phase with 2 months of flexible dose titration to the MTD followed by a period of stable treatment, and will continue the language intervention throughout. A post-intervention follow-up visit will be conducted one month after the final assessment visit of the trial.

Researchers will compare overall weighted communication score in the AFQ056 and placebo groups, after 6 months of treatment in combination with an intensive standardized parent-implemented language learning intervention. This is meant to serve as a marker of drug effect on neural plasticity, the core problem in the disorder. Further assessments will also be compared between groups to determine changes in language, cognitive, and adaptive functioning.

ELIGIBILITY:
Inclusion Criteria

1. Age 32 months to 6 years inclusive at Screening (visit 1).
2. Has an FMR1 full mutation.

   **Note Presence of mosaicism is allowed
3. DQ<75 calculated from the Mullen Scales of Early Learning at time of screening.
4. Parent or legal guardian is available and able to communicate well with the investigator, comply with study requirements and provide written informed consent.

   **Note**The Parent or legal guardian who will be signing consent form, should be the individual administering the language intervention
5. English is the primary language spoken in the home and the subject's first language is English.
6. Meet criteria indicating evidence of intentional communication based on parent interview via a communication eligibility screening tool.

   **Note** On the Eligibility Screening Tool - Communication, the child must have at time of screening:
   1. Section 1: Answer of YES; the child uses at least 5 spoken words to label items on a daily basis.

      OR
   2. Section 2: At least 3 YES answers to items 1-10 if child does not have at least 5 spoken words.
7. Produces 3 or more intentional acts of communication on the structured portion of the Weighted Communication play sample at time of screening.

   **Note: subjects are permitted to use augmentative communication devices throughout the study if the device is the subject's primary form of communication and the device has been prescribed for the subject by an SLP.
8. Stable behavioral and other therapy regimen for 30 days prior to screening.

   **Note: Patients will be allowed to continue their standard of care therapies throughout the trial but these will not be changed during the placebo lead in or placebo controlled portion of the trial, outside of the standard changes occurring from school schedules.
9. Stable dosing of all concurrent psychotropic medications except stimulants for at least 60 days prior to screening. Due to the very short half-life of stimulants (specifically methylphenidate and amphetamine variants), a stable regimen of these medications is required for 2 weeks only.

   * Note** Medications impacting GABA, glutamate and/or mGluR5 pathway receptors are exclusionary and not permitted during study participation. Additionally, stimulant regimens may include combinations of short- and long-acting forms and may be taken with different timing or dosing on different days of the week (e.g. Doses may be skipped on weekends or days off school and extra doses may be given some days for therapy sessions later in the day). The intent is to keep the doses and regimen being used at the time of screening consistent during the trial even if there is some variation in how the medication is taken on different days.Use of CBD oil or hemp based substances legal for sale over the internet are allowed provided that the dosing regimen has been consistent for at least 60 days prior to screening and will remain the same throughout the trial.

Exclusion Criteria

1. Use of medications impacting GABA, glutamate and/or mGluR5 pathway receptors or transmission.

   * Note** Treatment with acamprosate, amantadine, budipine, carbetocin, cycloserine, dextromethorphan, felbamate, ketamine, lithium, minocycline, memantine, oxytocin, remacemide, racemic baclofen, riluzole, fycampa, investigational mGluR5 medications, and/or statins are exclusionary.
   * Note** Lithium taken as a dietary supplement is permitted if the dose is less than 5mg/day. A 5mg/day dose is the recommended dietary intake level, and therefore is not considered to be therapeutic. Lithium dosage must remain the same throughout the duration of the trial and documented in the concomitant medication log.
2. Unstable seizure disorder as defined by any seizure in the 6 months prior to the screening visit, and/or any change in anti-convulsant drug dosing in the 60 days prior to screening.

   **Note** Use of levetiracetam and oxcarbazepine are among permitted anticonvulsants.
3. Use of any other investigational drug at the time of enrollment or within 30 days or 5 half-lives (whichever is longer) of the investigational drug prior to screening until end of study visits (or longer if required by local regulations).
4. History of hypersensitivity to AFQ056 or any mGluR antagonist.
5. History or presence of any clinically significant disease of any major system organ class, within the past 2 years prior to screening including but not limited to neurological, cardiovascular, endocrine, metabolic, renal, or gastrointestinal disorders. This does not include typical features of FXS such as psychological symptoms or history of epileptic seizures.
6. Significant acute illness that did not completely resolve at least four weeks prior to the Screening visit.
7. Abnormal laboratory values at screening that are in the opinion of the investigator are clinically significant and may jeopardize the safety of the study subject.
8. Use of (or use within at least 5 half-lives before dosing) concomitant medications that are strong/moderate inhibitors or inducers of CYP1A1/2, CYP2C9/19 or CYP3A4 (see Appendix B).
9. Subjects who are, in the opinion of the investigator, unable to comply with the requirements of the study.
10. Presence of immunodeficiency diseases at the time of screening, based on medical history, including a positive HIV test result.
11. History of a positive Hepatitis B surface antigen (HBsAg) or Hepatitis C result at time of screening.
12. History or presence of suicidal thoughts and/or suicide attempts.

Ages: 32 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Berry-Kravis, MD, PhD, Principal Investigator — Rush University Medical Center
Locations (14):
- United States (14):
  - Univeristy of California - Davis, Davis, California
  - Children's Hospital of Colorado, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - St Louis Children's Hospital (Washington University School of Medicine), St Louis, Missouri
  - Columbia University - New York Presbyterian, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Derived] Protic D, Breeze E, Mendoza G, Zafarullah M, Abbeduto L, Hagerman R, Coffey C, Cudkowicz M, Durbin-Johnson B, Ashwood P, Berry-Kravis E, Erickson CA, Filipink R, Gropman A, Lehwald L, Maxwell-Horn A, Morris S, Bennett AP, Prock L, Talboy A, Tartaglia N, Veenstra-VanderWeele J, Tassone F. Negative effect of treatment with mGluR5 negative allosteric modulator AFQ056 on blood biomarkers in young individuals with Fragile X syndrome. SAGE Open Med. 2024 Sep 29;12:20503121241282401. doi: 10.1177/20503121241282401. eCollection 2024. PMID 39483619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It is expected that recruitment/enrollment will occur over 18 months. Enrollment must end at the end of February 2020 due to study drug expiration at the end of August 2021.
Pre-assignment Details: Prior to randomization, there will be a 4-month single-blind placebo lead in after screening assessments during which subjects will have therapy treatments as usual to control for the effects of the language intervention. The placebo lead-in will also control for placebo effects which are prominent in clinical trials in FXS.
Groups:
- Placebo Lead-In: Children with FXS were seen for a screening visit and if they met entry criteria, they began a single-blind 4-month placebo lead-in period prior to randomization during which they received their therapy treatments as usual, with no language intervention.
- Double-Blind Placebo, Then Open-Label AFQ056: Double-Blind Placebo Period: After a 4-month single-blind placebo lead-in period, subjects with FXS were randomized to receive a placebo suspension by mouth twice per day in an 8 month double-blind treatment period.
  During the double-blind treatment period, dose titration to maximum tolerated dose of matching placebo occurred over 7 weeks. After 7 weeks, the dose was fixed, and at the 2 month visit, the intensive language intervention was initiated. Subjects continued the language intervention while remaining on placebo for the next 6 months.
  Safety and efficacy assessments were performed throughout.
  Open-Label Period: After 8 months of treatment in the placebo-controlled phase, all subjects had assessments completed and were given the opportunity to enter the open-label extension (OLE) in which all subjects received AFQ056. The OLE began with 2 months of flexible dose titration to each subject's maximum tolerated dose followed by a period of stable treatment. Subjects also continued the language intervention through the extension phase.
  The total duration of the OLE depended on when the subject was enrolled into the study and ranged from no open label to 8 months.
- Double-Blind AFQ056, Then Open-Label AFQ056: Double-Blind Placebo Period: After a 4-month single-blind placebo lead-in period, subjects with FXS were randomized to receive AFQ056 suspension by mouth twice per day in an 8 month double-blind treatment period.
  During the double-blind treatment period, subjects in the AFQ056 treatment group began with a dose of 25 mg AFQ056 twice per day and titrated to their maximum tolerated dose over the course of 7 weeks. After 7 weeks the dose was fixed, and at the 2 month visit, the intensive language intervention was initiated. Subjects continued the language intervention while remaining on a stable dose of AFQ056 (ranging from 12.5 mg BID to 100 mg BID), for the next 6 months.
  Safety and efficacy assessments were performed throughout.
  Open-Label Period: After 8 months of treatment in the placebo-controlled phase, all subjects had assessments completed and were given the opportunity to enter the open-label extension (OLE) in which all subjects received AFQ056. The OLE began with 2 months of flexible dose titration to each subject's maximum tolerated dose followed by a period of stable treatment. Subjects also continued the language intervention through the extension phase.
  The total duration of the OLE depended on when the subject was enrolled into the study and ranged from no open label to 8 months.
Period: Placebo Lead-In Period
Arm/Group | Placebo Lead-In | Double-Blind Placebo, Then Open-Label AFQ056 | Double-Blind AFQ056, Then Open-Label AFQ056
Started | 110 | 0 | 0
Completed | 99 | 0 | 0
Not Completed | 11 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Subject Ineligible | 6 | 0 | 0
Not completed — Subject Screen Fail | 4 | 0 | 0
Period: Placebo-Controlled Period
Arm/Group | Placebo Lead-In | Double-Blind Placebo, Then Open-Label AFQ056 | Double-Blind AFQ056, Then Open-Label AFQ056
Started | 0 | 49 | 50
Completed | 0 | 46 | 43
Not Completed | 0 | 3 | 7
Not completed — Withdrawal by Subject | 0 | 3 | 5
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Period: Open-Label Extension (OLE) Period
Arm/Group | Placebo Lead-In | Double-Blind Placebo, Then Open-Label AFQ056 | Double-Blind AFQ056, Then Open-Label AFQ056
Started | 0 | 46 | 43
Completed | 0 | 37 | 39
Not Completed | 0 | 9 | 4
Not completed — Withdrawal by Subject | 0 | 5 | 2
Not completed — Study Drug Expiration | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo Comparator: Double-Blind Placebo With Language Intervention: After a 4-month single-blind placebo lead-in period, subjects with FXS were randomized to receive a placebo suspension by mouth twice per day in an 8 month double-blind treatment period.
  During the double-blind treatment period, dose titration to maximum tolerated dose of matching placebo occurred over 7 weeks. After 7 weeks, the dose was fixed, and at the 2 month visit, the intensive language intervention was initiated. Subjects continued the language intervention while remaining on placebo for the next 6 months.
  Safety and efficacy assessments were performed throughout.
- Experimental: Double-Blind AFQ056 With Language Intervention: After a 4-month single-blind placebo lead-in period, subjects with FXS were randomized to receive AFQ056 suspension by mouth twice per day in an 8 month double-blind treatment period.
  During the double-blind treatment period, subjects in the AFQ056 treatment group began with a dose of 25 mg AFQ056 twice per day and titrated to their maximum tolerated dose over the course of 7 weeks. After 7 weeks the dose was fixed, and at the 2 month visit, the intensive language intervention was initiated. Subjects continued the language intervention while remaining on a stable dose of AFQ056 (ranging from 12.5 mg BID to 100 mg BID), for the next 6 months.
  Safety and efficacy assessments were performed throughout.
- Total: Total of all reporting groups
Arm/Group | Placebo Comparator: Double-Blind Placebo With Language Intervention | Experimental: Double-Blind AFQ056 With Language Intervention | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.1 (1.4) | 5.3 (1.3) | 5.2 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 42 | 46 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 43 | 42 | 85
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 1 | 4
  White | 43 | 41 | 84
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 47 | 50 | 97
  China | 2 | 0 | 2
Weighted Child Intentional Communication Score [Mean (Standard Deviation); unit: score on a scale] — The Weighted Child Intentional Communication Score is coded from a 22 minute semi-structured examiner/child play session. The score reflects child initiated communication that involves the child's use of gestures, eye contact, vocalizations, and/or words and word combinations to communicate a message to a listener. Higher scores indicate more child-initiated communication. There is no maximum score.
  score on a scale | 282.8 (264.2) | 304.0 (270.2) | 293.2 (266.0)
Mullen Scales of Early Learning (MSEL) Developmental Quotient (DQ) [Mean (Standard Deviation); unit: units on a scale] — The MSEL measures performance over 5 subscales: gross motor, fine motor, visual reception, expressive language, and receptive language. Developmental age can be calculated by averaging the developmental age equivalents from 4 domains of the Mullen (visual reception, fine motor, receptive language, and expressive language). To calculate the developmental quotient (DQ), developmental age in months is divided by chronological age in months and multiplied by 100. DQ values can range from 1 to 70. A higher DQ indicates better performance on the MSEL.
  units on a scale | 45.4 (14.4) | 43.9 (16.3) | 44.6 (15.3)
Mullen Scales of Early Learning (MSEL) Expressive Language Subscore [Mean (Standard Deviation); unit: score on a scale] — The MSEL measures performance over 5 subscales including expressive language. The range of possible subscores for the expressive language domain is 1-50. A higher score indicates better performance / greater use of expressive language.
  score on a scale | 22.5 (10.0) | 23.2 (10.7) | 22.9 (10.3)
Vineland Adaptive Behavior Scale (Vineland-3) Composite Score [Mean (Standard Deviation); unit: score on a scale] — The Vineland-3 is an informant-based measure that is administered using a semi-structured interview format. The assessment provides standard scores in domains of communication, daily living skills, socialization, and motor skills. The Adaptive Behavior Composite (ABC) is yielded from these domain scores and provides an overall summary measure of adaptive functioning.The range of possible composite scores is 20-140 with a higher score indicating higher levels of adaptive functioning.
  score on a scale | 66.0 (10.3) | 64.0 (12.2) | 65.0 (11.3)
Vineland Adaptive Behavior Scale (Vineland-3) Communication Score [Mean (Standard Deviation); unit: score on a scale] — The communication domain of the Vineland-3 examines adaptive functioning in receptive, expressive, and written language.The range of possible subscores for the communication domain is 20-140 with a higher score indicating more advanced use of language.
  score on a scale | 61.2 (15.4) | 56.8 (19.1) | 59.0 (17.4)
Preschool Language Scale (PLS-5) Expressive Communication Score [Mean (Standard Deviation); unit: scores on a scale] — The PLS-5 is a comprehensive developmental language assessment that requires the child to point to or verbally respond to items. One domain that is evaluated using this assessment is expressive language. Higher scores represent greater use of expressive communication. It is difficult to specify an upper bound on the score, because there is no clear expectation of a limit on the number of times a child can communicate unless one sets it artificially (e.g., once per second in an 11-minute free play). The lower bound is zero for a child who produces no communication acts.
  scores on a scale | 28.8 (9.9) | 29.7 (10.7) | 29.2 (10.3)
MacArthur-Bates Communicative Development Inventory (CDI) Number of Spoken Words [Mean (Standard Deviation); unit: words] — The MacArthur-Bates CDI is a parent interview that allows tracking of a child's progress in developing words, sentences, and more complex language. The assessment consists of two parts including "Words Children Use," a 680-word vocabulary checklist in which the parent indicates those vocabulary words the child regularly produces in spoken language, and "Sentences and Grammar" an assessment of several aspects of grammar and word endings. The MacArthur-Bates CDI number of spoken words (raw scale) will be recorded with higher scores indicating more words used / greater language development.
  words | 262.8 (231.4) | 305.6 (253.3) | 284.2 (242.3)
Clinical Global Impression - Improvement: Overall Function [Count of Participants; unit: Participants] — The Overall Function CGI-I considers all areas of function including cognition, adaptive behavior, and maladaptive behavior and requires the clinician to rate how much the study participant's overall function has improved or worsened relative to a baseline state. The CGI-I is a 7-point scale that ranges from very much improved (1) to very much worse (7).
  The CGI-I at baseline was completed relative to overall function at screening.
  Participants
    Much/very much improved | 4 | 0 | 4
    Minimally improved | 4 | 11 | 15
    No change | 37 | 35 | 72
    Minimally worse | 3 | 4 | 7
    Much/very much worse | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Weighted Child Intentional Communication Score
Description: The Weighted Child Intentional Communication Score is derived from a 22 minute semi-structured examiner/child play session. Structured and unstructured component scores are found by multiplying each intentional communication act by the following weights: nonverbal = 1; single symbol = 2; and multiple symbols = 3. The two scores are summed together to obtain the total. Higher scores indicate more child-initiated communication. There is no maximum score.
  The scale was administered at Baseline, Month 2, Month 4, Month 6, and Month 8. A composite score representing the average of the estimated change scores calculated at months 2, 4, 6, and 8 was recorded. A higher least squares mean value indicates a greater increase in WCS score from baseline.
Time Frame: Baseline through Month 8
Population: Comparison of WCS from baseline and from month 8 visit (end of double-blind period) in both AFQ056 & Language Intervention and Placebo & Language Intervention groups.
Measure: Least Squares Mean (90% Confidence Interval); unit: log10(scores on a scale)
Groups:
- Placebo Comparator: Double-Blind Placebo With Language Intervention: Randomized to receive AFQ056-matched placebo twice per day in conjunction with the language intervention during the double-blind period.
- Experimental: Double-Blind AFQ056 With Language Intervention: Randomized to receive AFQ056 twice per day in conjunction with the language intervention during the double-blind period. Subjects will take between 25-100 mg BID orally. Dose will depend on individual patient max tolerance.
Arm/Group | Placebo Comparator: Double-Blind Placebo With Language Intervention | Experimental: Double-Blind AFQ056 With Language Intervention
Number analyzed (Participants) | 49 | 50
log10(scores on a scale) | 0.14 [0.05 to 0.22] | 0.04 [-0.05 to 0.12]
Statistical Analysis 1: Comparison: Placebo Comparator: Double-Blind Placebo With Language Intervention vs Experimental: Double-Blind AFQ056 With Language Intervention; Test type: Superiority; p = 0.1587, Mixed Models Analysis; Slope = -0.1, 90% CI 2-sided [-0.22 to 0.02]

2. Secondary Outcome: Change in Mullen Scales of Early Learning (MSEL) Developmental Quotient (DQ)
Description: Mullen Scales of Early Learning (MSEL) Developmental Quotient (DQ) is calculated by averaging the developmental age equivalents from 4 domains of the Mullen (visual reception, fine motor, receptive language, and expressive language) to find developmental age in months, dividing by chronological age in months, then multiplying by 100. DQ can range from 1 to 70. A higher DQ indicates better performance on the MSEL.
  The MSEL was administered at Baseline, Month 2, and Month 8. A composite score representing the average of the estimated change scores calculated at month 2 and month 8 was recorded. A negative least squares mean indicates a net decrease in DQs over time. A more negative least squares mean indicates a larger negative change in DQs over time.
Time Frame: Baseline through Month 8
Population: Comparison of DQ from baseline and from month 8 visit (end of double-blind period) in both AFQ056 & Language Intervention and Placebo & Language Intervention groups.
Measure: Least Squares Mean (90% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo Comparator: Double-Blind Placebo With Language Intervention | Experimental: Double-Blind AFQ056 With Language Intervention
Number analyzed (Participants) | 49 | 50
scores on a scale | -0.7 [-1.90 to 0.50] | -2.35 [-3.55 to -1.16]
Statistical Analysis 1: Comparison: Placebo Comparator: Double-Blind Placebo With Language Intervention vs Experimental: Double-Blind AFQ056 With Language Intervention; Test type: Superiority; p = 0.1054, Mixed Models Analysis; Slope = -1.66, 90% CI 2-sided [-3.34 to 0.03]

3. Secondary Outcome: Change in Mullen Scales of Early Learning (MSEL) Expressive Language Subscore
Description: The MSEL measures performance over 5 subscales including expressive language. The range of possible subscores for the expressive language domain is 1-50. A higher score indicates better performance / greater use of expressive language
  The MSEL was administered at Baseline, Month 2, and Month 8. A composite score representing the average of the estimated change scores calculated at month 2 and month 8 was recorded. A positive least squares mean indicates a net positive change in expressive language scores over time. A higher least squares mean indicates a larger change in expressive language scores over time.
Time Frame: Baseline through Month 8
Population: Comparison of MSEL expressive language subscore from baseline and from month 8 visit (end of double-blind period) in both AFQ056 & Language Intervention and Placebo & Language Intervention groups.
Measure: Least Squares Mean (90% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo Comparator: Double-Blind Placebo With Language Intervention | Experimental: Double-Blind AFQ056 With Language Intervention
Number analyzed (Participants) | 49 | 50
scores on a scale | 1.99 [1.19 to 2.79] | 1.32 [0.52 to 2.11]
Statistical Analysis 1: Comparison: Placebo Comparator: Double-Blind Placebo With Language Intervention vs Experimental: Double-Blind AFQ056 With Language Intervention; Test type: Superiority; p = 0.32, Mixed Models Analysis; Slope = -0.67, 90% CI 2-sided [-1.79 to 0.45]

4. Secondary Outcome: Change in Vineland Adaptive Behavior Scale (Vineland-3) Composite Score
Description: The Vineland-3 composite score is yielded from the subject's level of adaptive functioning in the domains of communication, daily living skills, socialization, and motor skills. The range of possible composite scores is 20-140 with a higher score indicating higher levels of adaptive functioning.
  The Vineland-3 was administered at Baseline, Month 2, Month 4, Month 6, and Month 8. A composite score representing the average of the estimated change scores calculated at months 2, 4, 6, and 8 was recorded. A positive least squares mean indicates a net increase in composite score over time. A higher least squares mean indicates a greater change in composite score over time.
Time Frame: Baseline through Month 8
Population: Comparison of Vineland-3 Composite Score from baseline and from month 8 visit (end of double-blind period) in both AFQ056 & Language Intervention and Placebo & Language Intervention groups.
Measure: Least Squares Mean (90% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo Comparator: Double-Blind Placebo With Language Intervention | Experimental: Double-Blind AFQ056 With Language Intervention
Number analyzed (Participants) | 49 | 50
scores on a scale | 0.68 [-0.51 to 1.88] | 0.39 [-0.81 to 1.60]
Statistical Analysis 1: Comparison: Placebo Comparator: Double-Blind Placebo With Language Intervention vs Experimental: Double-Blind AFQ056 With Language Intervention; Test type: Superiority; p = 0.78, Mixed Models Analysis; Slope = -0.29, 90% CI 2-sided [-1.98 to 1.4]

5. Secondary Outcome: Change in Vineland Adaptive Behavior Scale (Vineland-3) Communication Subscore
Description: The communication domain of the Vineland-3 examines adaptive functioning in receptive, expressive, and written language. The range of possible subscores for the communication domain is 20-140 with a higher score indicating more advanced use of language.
  The Vineland-3 was administered at Baseline, Month 2, Month 4, Month 6, and Month 8. A composite score representing the average of the estimated change scores calculated at months 2, 4, 6, and 8 was recorded. A positive least squares mean indicates a net increase in communication score over time. A higher least squares mean indicates a greater change in communication score over time.
Time Frame: Baseline and Month 8
Population: Comparison of Vineland-3 Communication Subscore from baseline and from month 8 visit (end of double-blind period) in both AFQ056 & Language Intervention and Placebo & Language Intervention groups.
Measure: Least Squares Mean (90% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo Comparator: Double-Blind Placebo With Language Intervention | Experimental: Double-Blind AFQ056 With Language Intervention
Number analyzed (Participants) | 49 | 50
scores on a scale | 0.54 [-0.97 to 2.05] | 0.63 [-0.90 to 2.16]
Statistical Analysis 1: Comparison: Placebo Comparator: Double-Blind Placebo With Language Intervention vs Experimental: Double-Blind AFQ056 With Language Intervention; Test type: Superiority; p = 0.94, Mixed Models Analysis; Slope = 0.1, 90% CI 2-sided [-2.05 to 2.24]

6. Secondary Outcome: Change in Preschool Language Scale (PLS-5) Expressive Communication Score
Description: The PLS-5 is a comprehensive developmental language assessment that requires the child to point to or verbally respond to items. Raw scores for expressive language were collected from this test. It is difficult to specify an upper bound on the score, because there is no clear expectation of a limit on the number of times a child can communicate unless one sets it artificially (e.g., once per second in an 11-minute free play). The lower bound is zero for a child who produces no communication acts.
  The PLS-5 was administered at Baseline, Month 2, and Month 8. A composite score representing the average of the estimated change scores calculated at month 2 and month 8 was recorded. A higher least squares mean indicates a larger change in PLS-5 communication score over 8 months.
Time Frame: Baseline and Month 8
Population: Comparison of PLS-5 expressive communication scores from baseline and from month 8 visit (end of double-blind period) in both AFQ056 & Language Intervention and Placebo & Language Intervention groups.
Measure: Least Squares Mean (90% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo Comparator: Double-Blind Placebo With Language Intervention | Experimental: Double-Blind AFQ056 With Language Intervention
Number analyzed (Participants) | 49 | 50
scores on a scale | 1.78 [1.10 to 2.46] | 0.93 [0.25 to 1.60]
Statistical Analysis 1: Comparison: Placebo Comparator: Double-Blind Placebo With Language Intervention vs Experimental: Double-Blind AFQ056 With Language Intervention; Test type: Superiority; p = 0.1428, Mixed Models Analysis; Slope = -0.85, 90% CI 2-sided [-1.81 to 0.11]

7. Secondary Outcome: MacArthur-Bates Communicative Development Inventory (CDI) Number of Spoken Words
Description: The MacArthur-Bates CDI is a parent interview that allows tracking of a child's progress in developing words, sentences, and more complex language. The assessment consists of two parts including "Words Children Use," a 680-word vocabulary checklist in which the parent indicates those vocabulary words the child regularly produces in spoken language, and "Sentences and Grammar" an assessment of several aspects of grammar and word endings. The MacArthur-Bates CDI number of spoken words will be recorded with higher scores indicating more words used / greater language development at Month 8.
Time Frame: Month 8
Population: Number of words spoken at month 8 visit (end of double-blind period) in both AFQ056 & Language Intervention and Placebo & Language Intervention groups.
Measure: Median (Full Range); unit: Spoken Words
Arm/Group | Placebo Comparator: Double-Blind Placebo With Language Intervention | Experimental: Double-Blind AFQ056 With Language Intervention
Number analyzed (Participants) | 49 | 50
Spoken Words | 319 [0 to 677] | 413.5 [0 to 680]
Statistical Analysis 1: Comparison: Placebo Comparator: Double-Blind Placebo With Language Intervention vs Experimental: Double-Blind AFQ056 With Language Intervention; Test type: Superiority; p = 0.24, Mixed Models Analysis; Odds Ratio (OR) = 0.9462, 90% CI 2-sided [0.8764 to 1.0215]

8. Secondary Outcome: Number of Participants With a Positive Response as Defined by Improvement in Clinical Global Impression - Improvement (CGI-I) Overall Function Scores
Description: Completion of the CGI-I requires the clinician to rate how much the study participant's illness has improved or worsened relative to a baseline state. For this study, two sets of CGI-I are administered at each applicable visit - one associated with Language/Communication and the other to Overall Function. The Overall Function CGI-I considers all areas of function including cognition, adaptive behavior, and maladaptive behavior. The CGI-I is a 7-point scale that includes the following ratings: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse.
  The CGI-I was rated at all study visits after screening. This measure shows the number of participants with positive CGI-I scores indicating perceived improvement at Month 8.
Time Frame: Month 8
Population: Patients with positive change in CGI-I scores from baseline to month 8 visit (end of double-blind period) in both AFQ056 & Language Intervention and Placebo & Language Intervention groups.
Measure: Number; unit: participants
Arm/Group | Placebo Comparator: Double-Blind Placebo With Language Intervention | Experimental: Double-Blind AFQ056 With Language Intervention
Number analyzed (Participants) | 49 | 50
participants | 10 | 8
Statistical Analysis 1: Comparison: Placebo Comparator: Double-Blind Placebo With Language Intervention vs Experimental: Double-Blind AFQ056 With Language Intervention; Test type: Superiority; p = 0.92, Mixed Models Analysis; Odds Ratio (OR) = 0.95, 90% CI 2-sided [0.4 to 2.27]

ADVERSE EVENTS:
Time Frame: Participants were monitored for AEs from the time they signed the consent until the final Study visit, up to 21 months. If an AE was ongoing or discovered at a subject's final Study visit, the AE was followed until resolution, or for a minimum of 30 days, whichever comes first.
Description: Adverse event review were done at all study visits, and during dose titration reviews. Safety monitoring was based on close observation of the child by the family. Children in the proposed age range who have developmental delay with a mental age of approximately 1-5 years are not be able to spontaneously communicate all (if any) side effects. Therefore, adverse event information was collected by querying caregivers about any differences in the child's behavior or wellbeing.
Groups:
- Placebo Lead-In Period: Children with FXS were seen for a screening visit and if they met entry criteria, they began a single-blind 4-month placebo lead-in period prior to randomization during which they received their therapy treatments as usual, with no language intervention.
- Double-Blind Period: Placebo With Language Intervention: Double-Blind Placebo Period: After a 4-month single-blind placebo lead-in period, subjects with FXS were randomized to receive a placebo suspension by mouth twice per day in an 8 month double-blind treatment period.
  During the double-blind treatment period, dose titration to maximum tolerated dose of matching placebo occurred over 7 weeks. After 7 weeks, the dose was fixed, and at the 2 month visit, the intensive language intervention was initiated. Subjects continued the language intervention while remaining on placebo for the next 6 months.
  Safety and efficacy assessments were performed throughout.
- Double-Blind Period: AFQ056 With Language Intervention: Double-Blind Placebo Period: After a 4-month single-blind placebo lead-in period, subjects with FXS were randomized to receive AFQ056 suspension by mouth twice per day in an 8 month double-blind treatment period.
  During the double-blind treatment period, subjects in the AFQ056 treatment group began with a dose of 25 mg AFQ056 twice per day and titrated to their maximum tolerated dose over the course of 7 weeks. After 7 weeks the dose was fixed, and at the 2 month visit, the intensive language intervention was initiated. Subjects continued the language intervention while remaining on a stable dose of AFQ056 (ranging from 12.5 mg BID to 100 mg BID), for the next 6 months.
  Safety and efficacy assessments were performed throughout.
- Open-Label Period: AFQ056 With Language Intervention: After 8 months of treatment in the placebo-controlled phase, all subjects had assessments completed and were given the opportunity to enter the open-label extension (OLE) in which all subjects received AFQ056. The OLE began with 2 months of flexible dose titration to each subject's maximum tolerated dose followed by a period of stable treatment. Subjects also continued the language intervention through the extension phase.
  The total duration of the OLE depended on when the subject was enrolled into the study and ranged from no open label to 8 months.
  The OLE included 46 patients who were previously assigned to placebo and 43 patients who were previously assigned to AFQ056.
Arm/Group | Placebo Lead-In Period | Double-Blind Period: Placebo With Language Intervention | Double-Blind Period: AFQ056 With Language Intervention | Open-Label Period: AFQ056 With Language Intervention
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/49 | 0/50 | 0/89
Serious Adverse Events (participants affected / at risk) | 1/110 | 1/49 | 0/50 | 1/89
Other Adverse Events (participants affected / at risk) | 65/110 | 44/49 | 45/50 | 76/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Lead-In Period (N=110) | Double-Blind Period: Placebo With Language Intervention (N=49) | Double-Blind Period: AFQ056 With Language Intervention (N=50) | Open-Label Period: AFQ056 With Language Intervention (N=89)
Atypical Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Croup Infectious (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Lead-In Period (N=110) | Double-Blind Period: Placebo With Language Intervention (N=49) | Double-Blind Period: AFQ056 With Language Intervention (N=50) | Open-Label Period: AFQ056 With Language Intervention (N=89)
Diarrhea (Gastrointestinal disorders) | 7 (8) | 3 (3) | 7 (8) | 10 (13)
Vomiting (Gastrointestinal disorders) | 9 (16) | 9 (9) | 4 (7) | 11 (17)
Pyrexia (General disorders) | 4 (4) | 1 (1) | 4 (5) | 5 (6)
Gastroenteritis (Infections and infestations) | 11 (12) | 7 (7) | 3 (3) | 6 (7)
Otitis Media (Infections and infestations) | 6 (7) | 9 (11) | 8 (11) | 8 (9)
Pharyngitis Streptococcal (Infections and infestations) | 4 (4) | 0 (0) | 3 (3) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 21 (24) | 17 (23) | 22 (37) | 41 (55)
Psychomotor Hyperactivity (Nervous system disorders) | 3 (3) | 10 (10) | 5 (5) | 25 (30)
Sensory Processing Disorder (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 5 (5)
Aggression (Psychiatric disorders) | 0 (0) | 3 (3) | 6 (6) | 7 (8)
Agitation (Psychiatric disorders) | 4 (4) | 8 (8) | 4 (5) | 5 (5)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (3) | 3 (3) | 10 (11)
Attention Deficit Hyperactivity Disorder (Psychiatric disorders) | 2 (2) | 3 (3) | 3 (3) | 7 (7)
Insomnia (Psychiatric disorders) | 7 (7) | 12 (14) | 17 (19) | 18 (20)
irritability (Psychiatric disorders) | 6 (6) | 7 (8) | 13 (13) | 13 (17)
Perseveration (Psychiatric disorders) | 1 (1) | 5 (5) | 3 (3) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 2 (2) | 6 (7) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 3 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT02920892/Prot_SAP_000.pdf